CLINICAL TRIAL: NCT02641483
Title: Afferent Stimulation to Evoke Recto-colonic Reflex for Colonic Motility
Brief Title: Stimulation for Colonic Motility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B1962-W
Record Dates: First submitted 2015-12-22; First posted 2015-12-29 (Estimated); Results first posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2022-11

CONDITIONS: Neurogenic Bowel Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Colonic Motility (Experimental): Study participants will act as their own controls, first providing data using their usual digital rectal stimulation intervention for bowel care, then providing data using electrical stimulation for bowel care.
  Interventions: Other: Electrical Rectal Stimulation

INTERVENTIONS:
Other: Electrical Rectal Stimulation — Electrical stimulation of the rectum will be applied to activate sensory afferent neurons of the rectum and evoke a recto-colonic reflex to improve colonic motility. This intervention will compared to individuals' usual mechanical intervention of digital rectal stimulation.

SUMMARY:
The investigators are testing the effect of electrical stimulation of the rectum on colonic motility. Most individuals with spinal cord injury develop neurogenic bowel dysfunction, which includes slowed colonic motility, which means that stools take longer than normal to pass through the colon. This slowed movement may result in chronic constipation and difficulty emptying the bowels. Individuals typically (without or without caregiver assistance) insert a gloved finger into the rectum and gently stretch it to improve colonic motility for a brief period to empty the bowels. The investigators hypothesize that electrically stimulating the rectum, instead of mechanically stretching it, will produce the same beneficial effect of improving colonic motility. Therefore, this study will compare the two methods. If electrical stimulation effectively improves colonic motility, then the investigator shall develop the approach as a therapeutic intervention in future studies.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed neurogenic bowel dysfunction and using digital rectal stimulation
* Neurologically stable
* Skeletally mature
* Suprasacral spinal cord injury, stroke, or multiple sclerosis
* At least 6 months post neurological injury or disease diagnosis

Exclusion Criteria:

* Active sepsis
* Open pressure sores on or around pelvis
* Significant colon trauma or colostomy
* History of autonomic dysreflexia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Bourbeau, PhD, Principal Investigator — Louis Stokes VA Medical Center, Cleveland, OH
Locations (2):
- United States (2):
  - Syracuse VA Medical Center, Syracuse, NY, Syracuse, New York
  - Louis Stokes VA Medical Center, Cleveland, OH, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Colonic Motility
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Colonic Motility
Number analyzed (Participants) | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Compare Changes in Number of Interventions Used to Complete Bowel Routine, Including Electrical Rectal Stimulation (Treatment) Versus Mechanical Rectal Distension (Control)
Description: Two interventions will be tested, including the clinical standard of digital rectal stimulation and a novel approach using electrical stimulation of rectal sensory afferents, to determine the effect on colonic pressure. Typically several bouts of digital rectal stimulation are required to achieve complete bowel emptying. We will compare the number of bouts of digital rectal stimulation (control) with electrical rectal stimulation (treatment) required to achieve complete bowel emptying.
Time Frame: 1 month
Measure: Median (Full Range); unit: bouts of stimulation
Arm/Group | Colonic Motility
Number analyzed (Participants) | 2
bouts of stimulation
  Control | 4 [4 to 5]
  Intervention | 1 [1 to 3]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for each study participant during their participation period, from enrollment to their completion of study activities, which was approximately 6 weeks for each study participant.
Arm/Group | Colonic Motility
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-03): https://cdn.clinicaltrials.gov/large-docs/83/NCT02641483/Prot_SAP_000.pdf